CLINICAL TRIAL: NCT05223439
Title: Investigation of Balance and Gait in Neuropathic Pain Due to Lumbar Disc Degeneration
Brief Title: Balance and Gait on Neuropathic Pain Due to Lumbar Disc Degeneration
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: KA21/489
Record Dates: First submitted 2022-01-21; First posted 2022-02-04 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; Gait Analysis; Spatio-Temporal Analysis; Foot Pressure Distribution
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals diagnosed with neuropathic pain due to lumbar disc degeneration: Individuals with neuropathic pain due to lumbar disc degeneration were included in this group.
- Individuals with lumbar disc degeneration but no neuropathic pain: Individuals without neuropathic pain due to lumbar disc degeneration were included in this group.
- Healthy Controls: Healthy individuals who did not have any problems that would affect gait were included.

SUMMARY:
Chronic lumbar neuropathic pain, characterized by pain, numbness, tingling and muscle weakness in the lower extremities, is one of the most common neuropathic pain syndromes. It is expected that balance and gait disturbances will occur as a result of motor and sensory problems in patients with neuropathic pain due to lumbar disc degeneration. However, as far as the investigators know, there is no study in the literature describing the effects of neuropathic pain due to lumbar disc degeneration on balance and gait. Therefore, the aim of our study; To examine the effects of neuropathic pain due to lumbar disc degeneration on balance and gait.

DETAILED DESCRIPTION:
Chronic lumbar neuropathic pain, characterized by pain, numbness, tingling and muscle weakness in the lower extremities, is one of the most common neuropathic pain syndromes. Since postural balance is controlled by sensory information, central processing, and neuromuscular responses, any change in proprioception due to prolonged neuropathic pain, asymmetrical load of the lower extremities, timing of dysfunctional muscle activation, sequencing, and asymmetry in foot pressure can alter postural balance. Solid evidence for the long-term effects of lumbar neuropathic pain on postural balance is lacking and needs to be addressed in people with lumbar disc degeneration. Gait problems are seen in patients with lumbar neuropathic pain and they walk more slowly than healthy individuals. However, it is not known to what extent neuropathic pain or neurological dysfunction due to disc degeneration affects gait. In the light of this information; It is expected that balance and gait disturbances will occur as a result of motor and sensory problems in patients with neuropathic pain due to lumbar disc degeneration. However, as far as the investigators know, there is no study in the literature describing the effects of neuropathic pain due to lumbar disc degeneration on balance and gait. Therefore, the aim of our study; To examine the effects of neuropathic pain due to lumbar disc degeneration on balance and gait.

ELIGIBILITY:
Inclusion criteria for individuals with neuropathic pain due to lumbar disc degeneration:

* Being between the ages of 40-70
* Taking 4 points or more from the Douleur Neuropathique en 4 questions (DN4) questionnaire
* Taking 12 points or more from the Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) scale

Inclusion criteria for individuals with lumbar disc degeneration but no neuropathic pain:

* Being between the ages of 40-70
* Taking below 4 points from the Douleur Neuropathique en 4 questions (DN4) questionnaire
* Taking below 12 points from the Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) scale

Inclusion criteria of healthy individuals in the study:

* Being between the ages of 40-70
* Have no pain (Taking 1 point or less according to the Visual Pain Scale)

Exclusion Criteria:

* Individuals with pain complaints of different etiology
* Individuals with neurological diseases that may cause central neuropathic pain such as stroke, head trauma, multiple sclerosis
* Individuals who have undergone orthopedic surgery in the last 6 months
* Individuals using any medication for neuropathic pain
* Individuals with chronic pain syndrome such as Fibromyalgia Syndrome

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with lumbar disc degeneration and healthy individuals will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
E-LINK FP3 Force Plate | Baseline
  Measuring the symmetrical weight distribution in the anterior-posterior and left-right axes, the system enables the assessment of the ability to maintain postural stability on a static surface. While the patient is standing on the force platform, determine which direction the balance has shifted.
KoreBalance Balance Evaluation System | Baseline
  The KoreBalance balance evaluation platform has a variable air pressure bag system and tilt sensor to monitor 360° horizontal and 20° vertical movements.
Gait Velocity | Baseline
  Zebris Rehawalk computerized gait evaluation system is used to assess the spatio-temporal characteristics of the gait. The system consists of a treadmill and a computer. While the computer automatically detects the patient's hip, knee, and ankle, measures an individual's foot pressure on the ground. For gait assessment, patients walk at their preferred comfortable walking speed.
Step Length | Baseline
  Zebris Rehawalk computerized gait assessment system is used to evaluate the spatio-temporal characteristics of gait and to perform kinetic-kinematic analysis.
Foot pressure distribution | Baseline
  The dynamic foot pressure distribution is analyzed with the pedobarography integrated into Zebris Rehawalk computerized gait assessment system. The system consists of a treadmill and a computer. While the computer automatically detects the patient's hip, knee, and ankle, measures an individual's foot pressure on the ground. For gait assessment, patients walk at their preferred comfortable walking speed.
Cadence | Baseline
  Zebris Rehawalk computerized gait evaluation system is used to assess the spatio-temporal characteristics of the gait. The system consists of a treadmill and a computer. While the computer automatically detects the patient's hip, knee, and ankle, measures an individual's foot pressure on the ground. For gait assessment, patients walk at their preferred comfortable walking speed.

OTHER OUTCOMES:
Douleur Neuropathique 4 Questions (DN4) | Baseline
  DN4 is a scale consisting of 10 questions evaluating neuropathic pain. Seven items are related to pain symptoms and three items include a clinical examination. The scale asks whether patients have burning, painful cold, electric shock, tingling, prickling, numbness, and itching. In addition, sensory changes in the patient are examined with cotton, pins, and brushing. While 1 point is given for each item in scoring, a score of 4 or more indicates the presence of neuropathic pain. Taking 4 points or more from the DN4 is one of the criteria for identifying neuropathic pain in the study.
Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) | Baseline
  The LANSS is a validated questionnaire that consists of 7 items, can distinguish neuropathic pain from nociceptive pain, and is easy to score in clinical settings. The first part of the scale consists of 5 items questioning the pain symptoms and answered as yes or no. The patient is asked to think about the pain he or she has felt during the past week. In the second part, the presence of allodynia and the sharp-blunt threshold value is evaluated by sensory examination. The questionnaire is calculated between 0-24 points. Twelve points and above indicates neuropathic pain. Taking below 12 points from the LANSS scale is one of the criteria for identifying neuropathic pain in the study.
Visual Analog Scale (VAS) | Baseline
  Visual Analog Scale is a scale that evaluates pain on a horizontal line. On the line, the left side indicates 'no pain' and the right side indicates 'the most severe pain imaginable. Healthy individuals are asked to mark a point on the line according to the severity of the pain they feel.
Brief Pain Inventory | Baseline
  This inventory includes the recording of the clinical information of the patients and the evaluation of their pain, and the pain, the severity of the pain, the character of the pain, the treatment methods applied against the pain, the results of these methods and their social-emotional effects are recorded.
Oswestry Disability Index | Baseline
  It is an index that measures the level of functional disability of individuals due to pain. It includes ten sub-headings: severity of pain, personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life and travel. Each question is scored between 0 and 5. Scores ranging from 0-50 are converted into a percentage value with a special formula according to the number of questions answered. The functional status worsens as the percentage increases.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Seçkinoğulları, MSc, Study Chair — Hacettepe University; Zeliha Özlem Yörük, Assoc. Prof., Study Chair — Baskent University; Sibel Kibar, Assoc. Prof., Study Chair — Atılım University; Ferdi Yavuz, Assoc.Prof., Study Chair — European University of Lefke; Kadriye Armutlu, Prof., Study Director — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara
  - Başkent University, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Nezari NH, Schneiders AG, Hendrick PA. Neurological examination of the peripheral nervous system to diagnose lumbar spinal disc herniation with suspected radiculopathy: a systematic review and meta-analysis. Spine J. 2013 Jun;13(6):657-74. doi: 10.1016/j.spinee.2013.02.007. Epub 2013 Mar 15. PMID 23499340
- [Background] Khoromi S, Patsalides A, Parada S, Salehi V, Meegan JM, Max MB. Topiramate in chronic lumbar radicular pain. J Pain. 2005 Dec;6(12):829-36. doi: 10.1016/j.jpain.2005.08.002. PMID 16326371
- [Background] Frost LR, Bijman M, Strzalkowski ND, Bent LR, Brown SH. Deficits in foot skin sensation are related to alterations in balance control in chronic low back patients experiencing clinical signs of lumbar nerve root impingement. Gait Posture. 2015 May;41(4):923-8. doi: 10.1016/j.gaitpost.2015.03.345. Epub 2015 Apr 3. PMID 25887249
- [Background] Bonab M, Colak TK, Toktas ZO, Konya D. Assessment of Spatiotemporal Gait Parameters in Patients with Lumbar Disc Herniation and Patients with Chronic Mechanical Low Back Pain. Turk Neurosurg. 2020;30(2):277-284. doi: 10.5137/1019-5149.JTN.27499-19.2. PMID 32091127